CLINICAL TRIAL: NCT04572971
Title: Reliability and Validity of iOS in IPF
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20/LO/0970
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a condition where scar tissue (called fibrosis) builds up in the lungs. It usually gets worse over time. Fibrosis causes the lungs to become stiff, and reduces the amount of oxygen that the lungs can take up. People with IPF complain of worsening breathlessness, which limits their day to day activities.

Lung function tests are breathing tests that measure how well the lungs are working, and are used by doctors to decide whether to start or stop medicines in people with IPF. However, people with IPF tell us that lung function tests require a lot of effort, can make them cough and feel very short of breath. About 1 in 5 people with IPF are unable to perform lung function results accurately.

Impulse oscillometry (iOS) is a new type of breathing test. It uses sound waves to measure the stiffness of the lung. The test is very quick (30 seconds), does not require any effort from the patient, and only requires a patient to breathe in their usual way. iOS has been used successfully in children who are unable to perform normal lung function tests.

The investigators will assess whether people with IPF can perform iOS tests accurately and to compare their experiences of having iOS tests with their experience of performing current lung function tests. The investigators will also compare whether there is a relationship between iOS tests and the information gathered from the tests currently used by doctors to measure the impact of IPF (lung function tests, exercise tests, lung scans and questionnaires that measure quality of life).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic pulmonary fibrosis made by specialist multidisciplinary team according to international standards
2. Able to provide written informed consent

Exclusion Criteria:

1. Contraindication to performing conventional lung function tests, e.g untreated TB, haemoptysis, pneumothorax, unstable cardiovascular status, recent eye, thoracic or abdominal surgery, thoracic, abdominal or cerebral aneurysm, acute illness (including diarrhoea and vomiting)
2. Unable to create seal on mouthpiece

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPF
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
iOS measurements of reactance | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield hospitals, London, Gb-lnd, United Kingdom

IPD SHARING:
Plan to Share IPD: No